CLINICAL TRIAL: NCT00702637
Title: Modafinil for the Treatment of Fatigue and Excessive Daytime Sleepiness in Individuals With Traumatic Brain Injury
Brief Title: Study of Modafinil to Treat Fatigue in Persons With Traumatic Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Alan Weintraub, MD, Craig Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H133A020510; R01
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Fatigue
Keywords: Traumatic Brain Injury; Fatigue; Modafinil; Somnolence
MeSH Terms: conditions — Fatigue; Brain Injuries, Traumatic; Sleepiness | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The purpose of this study is to determine whether Modafinil is effective in: (1) reducing fatigue and excessive daytime sleepiness (EDS) in individuals with Traumatic Brain Injury (TBI); and (2) improving cognitive function and quality of life in individuals with TBI.

DETAILED DESCRIPTION:
Background: An estimated 5.3 million Americans are living with a TBI-related disability today. These persons may face many issues, however, two chronic problems seem common to a strikingly large number of those who survive TBI: fatigue and EDS.

Need for Research: Modafinil has been shown to be useful for fatigue and sleepiness in patients with depression, multiple sclerosis, Parkinson's disease and individuals with EDS secondary to a variety of sleep disturbances. However, there has not been any controlled evaluation of Modafinil use for the treatment of individuals with TBI to date.

Current and Future Research Activity: Approximately 60 participants with post-TBI fatigue will be randomly assigned to two 10-week periods of taking either Modafinil or placebo. Participants taking Modafinil during the first 10 weeks will be switched to placebo for the second 10 weeks. Similarly, participants taking placebo during the first 10 weeks will be switched to Modafinil for the second 10 weeks. Outcomes relating to fatigue and EDS will be collected weekly throughout the study. Other outcomes (including general health, depression, and cognitive function) will be collected at the start of each period, 4 weeks into each period, and again at the end of each period. It is hypothesized that participants taking Modafinil will report significantly less fatigue and EDS, report significantly better general health and depression scores, and perform significantly better on tests of cognitive performance in comparison to participants taking placebo.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who sustained a TBI
* were discharged from Craig Hospital following initial rehabilitation
* are at least one year post-injury
* have disabling symptoms of fatigue and/or EDS which compromise their ability to function optimally
* (if female) are surgically sterile, two years post-menopausal, or if of childbearing potential, are using a medially acceptable method of birth control and agree to continue use of this method for the duration of the study

Exclusion Criteria:

* Individuals who have Neurologic and/or neuropsychiatric difficulties and/or deficits which will obscure the evaluation of this medication's effectiveness -
* have a diagnosis of other likely causes of EDS
* have concurrent medication use and/or clinically significant systemic disease that may cause fatigue and/or diminished arousal
* have epilepsy
* currently use of any anti-epileptic medications or Warfarin
* have cardiovascular disease or risks
* have severe renal or hepatic impairment
* have significant psychiatric or behavioral disturbance which would obscure the evaluation of medication effectiveness
* are a pregnant or lactating female

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-10; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Self report of fatigue
Self report of EDS
Data collected at baseline, 4 weeks, and 10 weeks (for both phases of crossover study)

SECONDARY OUTCOMES:
Self report of general health
Self report of depressive symptomatology
Performance on tests of cognitive functioning
Data collected at baseline, 4 weeks, and 10 weeks (for both phases of crossover study)